CLINICAL TRIAL: NCT02337153
Title: Study of Validation of Measurements of the Movement of Stiff Treated Teeth and Orthodontic Corticotomy
Brief Title: Ankylosed Teeth Treatment by Bone Orthodontic Treatment
Acronym: OBS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Firm Orthodontics - Mauguio - French (Unknown); Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Other Study IDs: 9367
Record Dates: First submitted 2014-12-31; First posted 2015-01-13 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Ankylosed Teeth
Keywords: Orthodontique Bone Stretching
MeSH Terms: conditions — Tooth Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Codify the treatment of teeth by stiff Corticotomy technique. Evaluate the duration of treatment and tooth movement.

DETAILED DESCRIPTION:
Codify the treatment of teeth by stiff Corticotomy technique. Evaluate the duration of treatment and tooth movement.

During treatment the teeth by stiff Corticotomy, millimeter measurements are performed on a cohort of patients with this pathology. These measures take place during normal clinical phases and on all media such as, plaster models, photographs and radiological examinations performed at the beginning, during and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient in need of orthodontic treatment and presenting one or more teeth stiff
* Can meet the requirement of orthodontic treatment (attendance, quality of brushing)
* Showing no indication against General Surgery

Exclusion Criteria:

* A patient against indication for orthodontic treatment : Root resorption of teeth adjacent to stiff teeth, Dental anchoring Deficiency by multiple agenesis or agenesis of the adjacent teeth to teeth stiff, Loss of periodontal support or active periodontal disease
* A patient against indication to treatment with Corticotomy : General Pathology against indicating surgery, Proximity root with no possibility of improvement orthodontic preparation
* Inability to maintain a good level of oral hygiene and good cooperation.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient in need of orthodontic treatment and presenting one or more teeth stiff
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-04-07 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the distal view of the tooth mesial to the stiff corner of the adjacent tooth | Before orthodontic preparation, At the end of the orthodontic preparation on the day of surgery, Then 7 days, 15 days, 21 days, 30 days, 45 days, 60 days from the date of Surgery, at the end of the treatment of ankylosed teeth
  Millimeter caliper measurements from the point of view of tooth distal to mesial stiff angle of the adjacent tooth during care for treatment corticotomy

SECONDARY OUTCOMES:
Change of the mesial angle of the ankylosed tooth to the distal (or mesial) angle of the adjacent tooth | Before orthodontic preparation, At the end of the orthodontic preparation on the day of surgery, Then 7 days, 15 days, 21 days, 30 days, 45 days, 60 days from the date of Surgery, at the end of the treatment of ankylosed teeth
  Millimeter caliper measurements from the mesial angle of the ankylosed tooth to the distal (or mesial) angle of the adjacent tooth during care for treatment corticotomy
Change of the incisal edge of ankylosed tooth to the Incisal edge of lower incisor, In occlusion | Before orthodontic preparation, At the end of the orthodontic preparation on the day of surgery, Then 7 days, 15 days, 21 days, 30 days, 45 days, 60 days from the date of Surgery, at the end of the treatment of ankylosed teeth
  Millimeter caliper measurements of the incisal edge of the ankylosed tooth incisal edge of lower incisor in occlusion during care for treatment
Change of free gingival margin of the ankylosed tooth to the gingival margin of the distal adjacent tooth | Before orthodontic preparation, At the end of the orthodontic preparation on the day of surgery, Then 7 days, 15 days, 21 days, 30 days, 45 days, 60 days from the date of Surgery, at the end of the treatment of ankylosed teeth
  Millimeter caliper measurements from free gingival margin of the ankylosed tooth to the gingival margin of the distal adjacent tooth during care for treatment corticotomy
Change of free gingival margin of the ankylosed tooth to the gingival margin of the mesial adjacent tooth | Before orthodontic preparation, At the end of the orthodontic preparation on the day of surgery, Then 7 days, 15 days, 21 days, 30 days, 45 days, 60 days from the date of Surgery, at the end of the treatment of ankylosed teeth
  Millimeter caliper measurements from free gingival margin of the ankylosed tooth to the gingival margin of the mesial adjacent tooth during care for treatment corticotomy

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BOUSQUET, MCU PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier - AHU CSERD, Montpellier, France